CLINICAL TRIAL: NCT06423768
Title: The fMRI in CardiaC arrEst With Uncertain Prognosis (FACE-UP) Study
Brief Title: fMRI in CardiaC arrEst With Uncertain Prognosis
Acronym: FACE-UP
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Samuel Snider, MD, MD, Brigham and Women's Hospital
Other Study IDs: 2024P000703
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to determine whether specific advanced MRI measures are associated with functional outcomes in patients who are comatose after cardiac arrest. The main question[s] it aims to answer are:

Aim 1: Determine if stimulus-based functional MRI (fMRI)-measured activations are independently associated with favorable neurological outcomes after cardiac arrest

Aim 2: Determine if resting state functional MRI (rs-fMRI)-measured functional network connectivity is independently associated with favorable neurological outcomes after cardiac arrest.

Aim 3: Determine if diffusion tensor imaging (DTI)-measured white matter integrity is associated with favorable neurological outcomes after cardiac arrest.

Participants will undergo advanced MRI sequences at time of clinical MRI, and will be followed for 6 months post-arrest.

DETAILED DESCRIPTION:
Our goal here is to determine whether advanced functional MRI and DTI sequences add actionable prognostic information relative to standard clinical MRI in patients who remain comatose after cardiac arrest. We plan the following specific analyses:

Aim 1: We will use logistic regression to measure the association between our primary outcome and fMRI BOLD response to (a) passive language stimuli, (b) motor imagery or (c) passive sensory stimuli, in a model with age, Glasgow Coma Scale (GCS) score at time of MRI, and presence of anoxic injury on clinical diffusion weighted MRI.

Aim 2: We will use logistic regression to measure the association between our primary outcome and default mode network resting state functional connectivity, in a model with age, Glasgow Coma Scale (GCS) score at time of MRI, and presence of anoxic injury on clinical diffusion weighted MRI.

Aim 3: We will use logistic regression to measure the association between our primary outcome and diffusion tensor imaging (DTI)-measured mean white matter fractional anisotropy, in a model with age, Glasgow Coma Scale (GCS) score at time of MRI, and presence of anoxic injury on clinical diffusion weighted MRI.

ELIGIBILITY:
Inclusion Criteria:

* survive of an in or out of hospital cardiac arrest

Exclusion Criteria:

* Drug overdose
* Opinion of medical team patient unlikely to survive more than 24 hours (severe concurrent medical illness, dilated and unreactive pupils, etc..)
* Following verbal commands (MD or RN note) once TTM is complete and normothermia is achieved (Day 2 or 3; Day of admission is Hospital Day 0). If no TTM is administered, this can be assessed on Hospital Day 2.
* Following verbal commands (study team assessment) at time of MRI
* Family planning to WLST at time of enrollment
* Non English speaker (okay if English not primary language, as long as they can understand it)
* Permanent Contraindication to MRI (some kind of implanted metal)
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who have survive a cardiac arrest but remain unresponsive after completion of targeted temperature management (TTM).
  We will enroll a separate sample of 15 healthy controls to provide a normative range for our advanced MRI imaging measures.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Cerebral Performance Category Score 1-2 | 6 months
  A standardized scale describing a patients overall level of independent function. Levels 1-2 reflect patients who are functionally independent in their iADLs.

SECONDARY OUTCOMES:
Cerebral Performance Category Score 1-3 | 2 weeks
  Any patient who has recovered consciousness (follows verbal commands), regardless of their disability level at 2-weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to post to openneuro.org